CLINICAL TRIAL: NCT05392673
Title: Comparative Analysis on Short-term Efficacies of Two Kinds of Artificai Liver Method in Treating Severe Hepatitis B.
Brief Title: Efficacy and Economic Evaluation of Nonbiological Artificial Liver Therapy in Acute-on-chronic Hepatitis B Liver Failure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202201022
Record Dates: First submitted 2022-05-09; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-03

CONDITIONS: Chronic-on-acute Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- comprehensive medical treatment (Experimental): All the 62 patients enrolled received comprehensive medical treatment after admission to the hospital, including anti-viral treatment, general supportive treatment, supplementation of blood products, such as albumin and plasma, and symptomatic treatment.
  Interventions: Other: KM-8800 plasma exchange device (Kuraray, Tokyo, Japan)
- PE(plasma exchange) (Experimental): In addition to comprehensive medical treatment, the PE groups were treated with PE or PE plus half-dose sequential PE. In the current study, PE was carried out using the KM-8800 plasma exchange device (Kuraray, Tokyo, Japan). The device was pre-flushed with 2000 mL of normal saline and 20 U/mL heparin dilution. And the blood pump speed was 100 to 120 mL/min and the plasma exchange speed was 25 to 30 mL/min. Before PE, calcium gluconate and diphenhydramine were routinely administrated to prevent an allergic reaction. For each time of plasma exchange,2800 mL fresh frozen plasma was administrated.
  Interventions: Other: KM-8800 plasma exchange device (Kuraray, Tokyo, Japan)
- DPMAS+half-dose sequential PE (Experimental): DPMAS with half-dose sequential PE was applied using the EC-40W plasma separator (Asahi Kasei Medical, Tokyo, Japan), BS330 bilirubin adsorption column (Jianfan Biotechnology, Zhuhai, China), and the neutral microporous adsorption resin HA330-Ⅱ (Jianfan Biotechnology). After the bilirubin adsorption and hemoperfusion treatment, sequential half-dose PE treatment begins. 1400 mL plasma replacement was conducted each time.
  Interventions: Other: KM-8800 plasma exchange device (Kuraray, Tokyo, Japan)

INTERVENTIONS:
Other: KM-8800 plasma exchange device (Kuraray, Tokyo, Japan) — Artificial liver scavenges inflammatory factors.
  Other Names: EC-40W plasma separator (Asahi Kasei Medical, Tokyo, Japan); BS330 bilirubin adsorption column (Jianfan Biotechnology, Zhuhai, China); The neutral microporous adsorption resin HA330-Ⅱ (Jianfan Biotechnology)

SUMMARY:
This was a non-blinded, prospective clinical study. From June 2020 to October 2021, 254 patients with HBV-ACLF were treated at the Department of Infectious Diseases, Xiangya Hospital, Central South University (Changsha, China). 186 patients who met the enrollment criteria were included in this study. Inclusion criteria were as follows: (1) aged 18-65 years old; (2) patients with ACLF caused by HBV infection; (3) meeting the diagnostic criteria for ACLF by the Asian Pacific Association for the Study of Liver (APASL).The exclusion criteria were as follows: (1) pregnancy or lactation; (2) previous liver transplantation; (3) hepatocellular carcinoma or other malignancy; (4) human immunodeficiency virus(HIV) infection or other immunocompromised states; (5) complicated with underlying diseases such as severe heart, respiratory, and blood system diseases. Based on the inclusion and exclusion criteria, the investigators randomly matched patients at a 1:1:1 ratio to three groups whose age, sex ratio, complication, and liver function were comparable: comprehensive medical treatment (Control group), PE group, and DPMAS plus half-dose sequential PE (DPMAS + PE group). As a result, 62 subjects per group were recruited into the study. This study was approved by the Clinical Research Ethics Committee of Xiangya Hospital, Central South University with informed content obtained from all participants (No. 202201022). The study protocol followed the principles of the Helsinki Declaration strictly.

All the 186 patients enrolled received comprehensive medical treatment after admission to the hospital, including anti-viral treatment, general supportive treatment, supplementation of blood products, such as albumin and plasma, and symptomatic treatment.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years old
* patients with ACLF caused by HBV infection
* meeting the diagnostic criteria for ACLF by the Asian Pacific Association for the Study of Liver.

Exclusion Criteria:

* pregnancy or lactation
* previous liver transplantation
* hepatocellular carcinoma or other malignancy
* human immunodeficiency virus(HIV) infection or other immunocompromised state
* complicated with underlying diseases such as severe heart, respiratory, and blood system diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with survival without liver transplantation | 90 days
Number of Participants with death | 90 days
Number of Participants with Liver transplantation | 90 days

SECONDARY OUTCOMES:
Progress of biochemical indexes | 90 days
  elevated bilirubin and transaminase

CONTACTS AND LOCATIONS:
Overall Officials: Wenting Peng, Principal Investigator — Xiangya Hospital of Central South University, Changsha, Hunan Province
Locations (1):
- Xiangya Hospital of Central South University, Changsha, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu T, Li J, Shao L, Xin J, Jiang L, Zhou Q, Shi D, Jiang J, Sun S, Jin L, Ye P, Yang L, Lu Y, Li T, Huang J, Xu X, Chen J, Hao S, Chen Y, Xin S, Gao Z, Duan Z, Han T, Wang Y, Gan J, Feng T, Pan C, Chen Y, Li H, Huang Y, Xie Q, Lin S, Li L, Li J; Chinese Group on the Study of Severe Hepatitis B (COSSH).. Development of diagnostic criteria and a prognostic score for hepatitis B virus-related acute-on-chronic liver failure. Gut. 2018 Dec;67(12):2181-2191. doi: 10.1136/gutjnl-2017-314641. Epub 2017 Sep 19. PMID 28928275
- [Result] Li H, Chen LY, Zhang NN, Li ST, Zeng B, Pavesi M, Amoros A, Mookerjee RP, Xia Q, Xue F, Ma X, Hua J, Sheng L, Qiu DK, Xie Q, Foster GR, Dusheiko G, Moreau R, Gines P, Arroyo V, Jalan R. Characteristics, Diagnosis and Prognosis of Acute-on-Chronic Liver Failure in Cirrhosis Associated to Hepatitis B. Sci Rep. 2016 May 5;6:25487. doi: 10.1038/srep25487. PMID 27146801
- [Result] Sarin SK, Choudhury A, Sharma MK, Maiwall R, Al Mahtab M, Rahman S, Saigal S, Saraf N, Soin AS, Devarbhavi H, Kim DJ, Dhiman RK, Duseja A, Taneja S, Eapen CE, Goel A, Ning Q, Chen T, Ma K, Duan Z, Yu C, Treeprasertsuk S, Hamid SS, Butt AS, Jafri W, Shukla A, Saraswat V, Tan SS, Sood A, Midha V, Goyal O, Ghazinyan H, Arora A, Hu J, Sahu M, Rao PN, Lee GH, Lim SG, Lesmana LA, Lesmana CR, Shah S, Prasad VGM, Payawal DA, Abbas Z, Dokmeci AK, Sollano JD, Carpio G, Shresta A, Lau GK, Fazal Karim M, Shiha G, Gani R, Kalista KF, Yuen MF, Alam S, Khanna R, Sood V, Lal BB, Pamecha V, Jindal A, Rajan V, Arora V, Yokosuka O, Niriella MA, Li H, Qi X, Tanaka A, Mochida S, Chaudhuri DR, Gane E, Win KM, Chen WT, Rela M, Kapoor D, Rastogi A, Kale P, Rastogi A, Sharma CB, Bajpai M, Singh V, Premkumar M, Maharashi S, Olithselvan A, Philips CA, Srivastava A, Yachha SK, Wani ZA, Thapa BR, Saraya A, Shalimar, Kumar A, Wadhawan M, Gupta S, Madan K, Sakhuja P, Vij V, Sharma BC, Garg H, Garg V, Kalal C, Anand L, Vyas T, Mathur RP, Kumar G, Jain P, Pasupuleti SSR, Chawla YK, Chowdhury A, Alam S, Song DS, Yang JM, Yoon EL; APASL ACLF Research Consortium (AARC) for APASL ACLF working Party.. Acute-on-chronic liver failure: consensus recommendations of the Asian Pacific association for the study of the liver (APASL): an update. Hepatol Int. 2019 Jul;13(4):353-390. doi: 10.1007/s12072-019-09946-3. Epub 2019 Jun 6. PMID 31172417
- [Result] Li LJ, Zhang YM, Liu XL, Du WB, Huang JR, Yang Q, Xu XW, Chen YM. Artificial liver support system in China: a review over the last 30 years. Ther Apher Dial. 2006 Apr;10(2):160-7. doi: 10.1111/j.1744-9987.2006.00358.x. PMID 16684218
- [Result] Karvellas CJ, Subramanian RM. Current Evidence for Extracorporeal Liver Support Systems in Acute Liver Failure and Acute-on-Chronic Liver Failure. Crit Care Clin. 2016 Jul;32(3):439-51. doi: 10.1016/j.ccc.2016.03.003. PMID 27339682
- [Result] Keklik M, Sivgin S, Kaynar L, Pala C, Solmaz M, Cetin M, Eser B, Unal A. Treatment with plasma exchange may serve benefical effect in patients with severe hyperbilirubinemia: a single center experience. Transfus Apher Sci. 2013 Jun;48(3):323-6. doi: 10.1016/j.transci.2013.04.009. Epub 2013 Apr 16. PMID 23602141
- [Result] Xu W, Li Y, Wang L, Gao H, Chen J, Yuan J, Ouyang Y, Gao Y, Li J, Li X, Peng L. Efficacy and safety of combination treatment of double plasma molecular adsorption system and low volume plasma exchange for patients with hepatitis B virus related acute-on-chronic liver failure: a multicentre randomised controlled clinical trial. BMJ Open. 2021 Dec 14;11(12):e047690. doi: 10.1136/bmjopen-2020-047690. PMID 34907041
- [Result] Guo X, Wu F, Guo W, Zhang J, Yang Y, Lu Y, Yin C, Fan H, Xu J, Liao M. Comparison of plasma exchange, double plasma molecular adsorption system, and their combination in treating acute-on-chronic liver failure. J Int Med Res. 2020 Jun;48(6):300060520932053. doi: 10.1177/0300060520932053. PMID 32552092